CLINICAL TRIAL: NCT07218055
Title: Assessment of Music Experiences in Navigating Depression (AMEND)
Brief Title: Assessment of Music Experiences in Navigating Depression Part 2
Acronym: AMEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Third Street Music School (Unknown)
Responsible Party: Principal Investigator, Joanne Loewy, Professor/Director, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STUDY-22-01609-CR004; STUDY-22-01609-CR004 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: Children's sadness; anxiety; fragility; music experiences in child assessment
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Ransom assignment to intervention or control across 6 month period-11 sessions
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomly assigned to treatment or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music (Experimental): Will receive assessment of music and 11 music therapy sessions as well as pretesting and f/u testing
  Interventions: Other: Music therapy
- Control (Sham Comparator): Will receive assessment of music pre-testing and follow up post testing
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — hourly weekly music therapy sessions
  Other Names: Verbal procession concert activity

SUMMARY:
This study is again looking at the use of music and music therapy experiences in navigating depression. The researchers will provide 11 sessions of music therapy and half will be followed by recitals at the Third Street School Music Settlement where the kids enrolled in our study will observe and interact with the performers and discuss and reflect on anxiety and performance and how sharing personal creativity affects them intra and interpersonally.

DETAILED DESCRIPTION:
The researchers will provide hourly weekly music therapy sessions and then go to the Third Street Music School and work with their kids and our kids providing insights and feedback. The researchers will test their depression (CDI) and Resilience (Connor Davidson)

ELIGIBILITY:
Inclusion Criteria:

- Must indicate depression -or symptoms thereof by parent in writing

Exclusion Criteria:

- none

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Conor-Davidson Resilience Scale | end of 6 months
  The Conor-Davidson Resilience Scale 10-item (Conor & Davidson, 2003, 2007) or CD-RISC10 is scale measuring the resilience of an individual. Each item is rated on a 5-point scale from 0 (not true at all) to 4 (True nearly all the time) with scoring from 0 to 40. The higher an individual scores, the greater their resilience. The lower an individual scores, the lower the individual's resilience.

SECONDARY OUTCOMES:
CDI2 or Children's Depression Inventory, Second Edition | end of 6 months
  The CDI2 is a self reported scale coming in two versions, CDI2 (28 items) and CDI2S (12 items). For this study, the CDI2S was chosen. Each item is rated on a 3-point scale from 0 to 2 with scoring from 0 to 24. 0 indicates no symptom, 1 indicates mild symptom, and 2 indicates definite symptom per item. The higher the total score, the stronger the indication for depression. Individuals who score from 0-12 indicate minimal to no depressive symptoms, individuals who score from 13-19 indicate mild depressive symptoms, and individuals who score 20 and above indicate moderate to severe depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Joanne V Loewy, D.A., LCAT, MT-BC, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to Shantelena.Mouzon@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included in the URL field below).
URL: https://www.mountsinai.org/locations/music-therapy